CLINICAL TRIAL: NCT04838223
Title: Neurosensory Abnormalities in SymptomAtic Ocular Surface Patients (NASA)
Acronym: NASA
Status: Suspended | Type: Observational
Why Stopped: PI is leaving insitution. This study is no longer active at TMC.
Sponsor: Tufts Medical Center (Other)
Collaborators: CooperVision International Limited (CVIL) (Industry); Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 00000319
Record Dates: First submitted 2020-08-19; First posted 2021-04-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye; Neuropathic Pain
MeSH Terms: conditions — Dry Eye Syndromes; Neuralgia | interventions — Single Person

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neuropathic Corneal Pain with Ocular Surface Discomfort: Participants diagnosed with neuropathic corneal pain with ocular surface discomfort
  Interventions: Other: Hyperosmolar Response; Other: Proparacaine Challenge Test; Other: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Optional; only for Contact Lens Wearers; Other: Ocular Pain Assessment Survey (OPAS); Other: Visual Analogue Questionnaire
- Neuropathic Corneal Pain with Dry Eye Disease: Participants diagnosed with dry eye disease and neuropathic corneal pain
  Interventions: Other: Hyperosmolar Response; Other: Proparacaine Challenge Test; Other: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Optional; only for Contact Lens Wearers; Other: Ocular Pain Assessment Survey (OPAS); Other: Visual Analogue Questionnaire
- NCP or Dry Eye in patients with ocular surface discomfort: Participants diagnosed with neuropathic corneal pain or with a neuropathic component of dry eye in patients with ocular surface discomfort
  Interventions: Other: Hyperosmolar Response; Other: Proparacaine Challenge Test; Other: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Optional; only for Contact Lens Wearers; Other: Ocular Pain Assessment Survey (OPAS); Other: Visual Analogue Questionnaire

INTERVENTIONS:
Other: Hyperosmolar Response — A single drop of hypertonic sodium chloride solution at room temperature will be instilled in each eye and change in pain/other symptoms after up to 90 seconds of application (to account for any initial irritation symptoms) will be observed.
Other: Proparacaine Challenge Test — A single drop of Proparacaine hydrochloride ophthalmic solution, (Alcaine®, 0.5%) will be used on each eye respectively and any change in pain/other symptoms will be noted after 90 seconds (to account for initial discomfort from the preservative in Proparacaine solution).
Other: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Optional; only for Contact Lens Wearers — The CLDEQ-8 is a validated eight-item scaled questionnaire developed to reflect the overall opinion of soft contact lenses.
Other: Ocular Pain Assessment Survey (OPAS) — Twenty seven-item quantitative questionnaire designed to provide an assessment of the symptoms and quality of life effect of ocular pain [18]. The 27 items of the OPAS questionnaire are graded on a scale of 0 to 10, or 10 to 100, where 0 indicates none and 10 or 100 indicate maximum.
Other: Visual Analogue Questionnaire — Symptoms of ocular comfort and dryness will be graded for each eye on a scale of 0-10, where 0=extremely uncomfortable, extremely dry and 10=excellent comfort, no dryness. An average rating will be provided for the morning, afternoon and evening.

SUMMARY:
This study is designed to measure how common nerve abnormalities are within a group of patients who feel discomfort within their eyes.

ELIGIBILITY:
Inclusion Criteria:

* Presents with ocular surface discomfort or for dry eye care
* Best corrected visual acuity of 20/40 or better in each eye
* Subject reported duration of symptoms of at least 3 months
* 100 subjects will be required to be habitual contact lens wearers as defined by use of contact lenses at least 5 hours per day at least 5 days per week for the last year.

Exclusion Criteria:

* Use of contact lenses on the day of the visit
* Pregnant or nursing
* Irregular corneas (e.g., ectatic disease, transplantation, or corneal dystrophies)
* Ocular surgery in the past 3 months
* Ocular infection in the past 3 months
* Active ocular allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,000 subjects will be enrolled for this study based on the above criteria:
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To establish the prevalence of neuropathic corneal pain in patients with ocular surface discomfort. | Day 1
  As measured by the percent of subjects who report increased ocular surface discomfort upon challenge with hyperosmolar saline.
To assess the overlap of neuropathic corneal pain with dry eye disease in patients in diseases that are currently thought to be mutually exclusive. | Day 1
  As measured by the percent of subjects who report ocular surface discomfort, and either do or do not exhibit signs of dry eye disease as defined by Tear Break Up Time, Schirmer's test, and staining, and have an increase in Visual Analog Scale score of more than 2 steps upon instillation of hypertonic saline.
To establish the prevalence of subtypes of patients with neuropathic corneal pain or with a neuropathic component of dry eye in patients with ocular surface discomfort. | Day 1
  As measured by the percent of subjects who report ocular surface discomfort, and have a decrease, partial decrease, or no change in Visual Analog Score score upon instillation of proparacaine.

SECONDARY OUTCOMES:
To assess the overlap of neuropathic corneal pain and contact lens discomfort. | 1 study visit
  Percent of contact lens wearers who report discomfort when wearing their contact lenses, and either do or do not exhibit signs of dry eye disease as defined by TBUT, Schirmer's test, and staining, and have an increase in VAS score of more than 2 steps upon instillation of hypertonic saline.
To establish the prevalence of anxiety/depression in patients with neuropathic corneal pain patients. | Day 1
  Percent of subjects who report increased ocular surface discomfort upon challenge with hyperosmolar saline and a history of anxiety/depression.
To assess for differences in in vivo confocal microscopy measures between dry eye disease patients and neuropathic corneal pain patients. | Day 1
  As measured by dendritic cell density, nerve fiber density, and microneuroma density
To assess for subtypes of neuropathic corneal pain differences in in vivo confocal microscopy measures between dry eye disease patients and neuropathic corneal pain patients. | Day 1
  As measured by dendritic cell density, nerve fiber density, and microneuroma density

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (16):
- United States (16):
  - Canyon City Eye Care, Azusa, California
  - Western University of Health Sciences, Pomona, California
  - University of California at San Francisco - Francis I Proctor Foundation, San Francisco, California
  - Bruce W. Carter VA Medical Center, Miami, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - Kannarr Eye Care, Pittsburg, Kansas
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Korb & Associates, Boston, Massachusetts
  - Midwest Vision Research Foundation at Prepose Vision Institute, St Louis, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Vita Eye Clinic, Shelby, North Carolina
  - SkyVision Centers, Westlake, Ohio
  - Hospital of the University of Pennsylvania (Scheie Eye Institute Perelman), Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No